CLINICAL TRIAL: NCT00156845
Title: A Phase 3, International, Multicenter, Open-Label, Dual-Injection, Echocardiographic Imaging and Safety Study in Patients With Suspected Ischemic Heart Disease Undergoing Diagnostic Coronary Angiography (Real-Time Assessment of Myocardial Perfusion With Echocardiography: RAMP 2)
Brief Title: Phase 3 Safety and Imaging Study of AI-700 in Patients With Suspected Coronary Artery Disease Undergoing Coronary Angiography
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Acusphere (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AI-700-33
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2006-07-14 (Estimated); Status verified 2006-07

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; ischemia; echocardiography; cardiac imaging; heart disease; myocardial contrast enhancement; myocardial perfusion; wall motion; ultrasound contrast agent
MeSH Terms: conditions — Coronary Artery Disease; Ischemia; Heart Diseases

INTERVENTIONS:
Procedure: AI-700 contrast-enhanced echocardiography

SUMMARY:
This study was designed to evaluate the ability of AI-700-enhanced rest-stress echocardiography to detect coronary artery disease (CAD) in patients with suspected ischemic heart disease who are indicated for coronary angiography.

DETAILED DESCRIPTION:
Assessment of myocardial perfusion has been demonstrated to provide both diagnostic and prognostic value to patients with ischemic heart disease by allowing the clinician to assess the hemodynamic significance of coronary artery disease (CAD). The primary objective of the clinical development program for AI-700 is to demonstrate the safety and efficacy of AI-700 as an intravenous ultrasound contrast agent in patients with suspected myocardial perfusion defects.

The patient population is comprised of patients being evaluated for inducible ischemia and indicated for coronary angiography. The primary study objective was to determine the accuracy, sensitivity, and specificity of AI-700-enhanced echocardiographic imaging for detecting CAD, using coronary angiography/left ventriculography (ANGIO/LVG) as the reference standard.

ELIGIBILITY:
Inclusion Criteria:

* Men and non-pregnant/non-lactating women with a history of typical or atypical chest pain (angina) who were 18 to 80 years of age and who had recently undergone coronary angiography or were scheduled for coronary angiography within 30 days after AI-700 administration were to be enrolled. Eligible patients must have also undergone SPECT for evaluation of CAD within 45 calendar days prior to AI-700 administration, or be scheduled for an "on-study" SPECT on the same day as AI-700 dosing or an "off-study" SPECT within 15 days following AI-700 dosing.

Exclusion Criteria:

* Study candidates who have had any of the following conditions were to be excluded from the study: any clinically unstable condition or major surgery within 7 days prior to AI-700 dosing; an acute MI; cerebrovascular accident or transient ischemic attack within 30 days prior to dosing; congestive heart failure graded as New York Heart Association Grade 4 within 3 months prior to dosing; significant left main CAD; previous coronary artery bypass graft; moderate to severe chronic obstructive pulmonary disease; or oxygen saturation < 90% at rest.
* Candidates with significant cardiovascular or pulmonary structural and/or functional abnormality, or in whom visualization of the left ventricle was not adequate for evaluation of cardiac function during the Exclusion ECHO, were to be ineligible to participate in the study.
* Patients who had a history of MI of non-CAD etiology or who exhibited new or changing ECG abnormalities at any time between Screening and AI-700 dosing were to be similarly excluded.
* Other exclusion criteria included: participation in an investigational drug/device study within 30 days prior to dosing (90 days in UK sites), non-seasonal asthma within the past 3 years or recent seasonal asthma requiring prescription medication, organ transplant or end-stage organ failure, and active seizure disorder.
* Candidates were to be excluded for uncontrolled atrial fibrillation, frequent premature ventricular or atrial contractions, history of prolonged QT/QTc, use of automatic implantable cardioverter/defibrillator or pacemaker, and any rhythm abnormality that had not been evaluated and treated by a specialist or for which current treatment did not ensure patient safety.
* Candidates who had used methylated xanthines within 24 hours of dosing were also to be excluded. Patients were also to be excluded if aminophylline, theophylline, or dipyridamole were contraindicated according to each agent's product labeling.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450
Dates: Start 2003-12; Study Completion 2006-06

PRIMARY OUTCOMES:
Accuracy, sensitivity, and specificity of AI-700 ECHO in assessing CAD
Safety of AI-700 administered IV to suspected CAD patients

CONTACTS AND LOCATIONS:
Locations (1):
- Acusphere, Inc., Watertown, Massachusetts, United States

REFERENCES:
- [Derived] Senior R, Monaghan M, Main ML, Zamorano JL, Tiemann K, Agati L, Weissman NJ, Klein AL, Marwick TH, Ahmad M, DeMaria AN, Zabalgoitia M, Becher H, Kaul S, Udelson JE, Wackers FJ, Walovitch RC, Picard MH; RAMP-1 and RAMP-2 Investigators. Detection of coronary artery disease with perfusion stress echocardiography using a novel ultrasound imaging agent: two Phase 3 international trials in comparison with radionuclide perfusion imaging. Eur J Echocardiogr. 2009 Jan;10(1):26-35. doi: 10.1093/ejechocard/jen321. PMID 19131498
- See also: Related Info — http://www.acusphere.com